CLINICAL TRIAL: NCT04409197
Title: Evaluation of Changes in Weight, Sleep, and Other Psycho-behavioural Parameters During Covid-19 Confinement in Subjects Monitored by the RNPC Network
Acronym: CO-RNPC
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: 38RC20.150
Record Dates: First submitted 2020-05-18; First posted 2020-06-01 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Comorbidities; Confinement; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During confinement, food intake can become compulsive, physical activity is significantly reduced, sleep is altered with exacerbated anxiety and stress levels and increased family violence. In some at-risk patients, mental health may even deteriorate. The temptation is great for all to take refuge in food or in front of screens. The main elements that can impact weight changes during this period of confinement are stress and anxiety, lack of physical activity, changes in eating habits, sleep disturbance and alcohol consumption.

The investigators wish to study the impact of confinement on pre-post confinement weight loss kinetics in adults included in weight reduction programs (RNPC).

ELIGIBILITY:
Inclusion Criteria:

* BMI > 25 kg/m² and/or waist circumference > 80 cm in women and 94 cm in men
* Persons registered in the RNPC program
* Be legally able to give consent after adequate information and submission of the information note
* Person affiliated to social security

Exclusion Criteria:

* Being unable to understand, follow objectives and methods due to cognition or language problems Subjects listed in articles L1121-5 à L1121-8: Pregnant women, feeding and parturient; subject under administrative or judicial control, persons who are protected under the act.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from patients enrolled in a Nutritional Psycho-Behavioural Re-education (RNPC) programme in one of the RNPC centres in France.
Sampling Method: Probability Sample
Enrollment: 4789 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-07-11 (Actual)

PRIMARY OUTCOMES:
Analyse the variation in weight loss kinetics before, during and after confinement in patients enrolled in a weight reduction programme (RNPC) in France | 3 months

SECONDARY OUTCOMES:
Define the effects of containment on the variation in the kinetics of anthropometric parameters other than weight | 3 months
  Change in waist circumference, blood pressure, percentage of lean, fluid and muscle mass before and after the confinement period
Evolution of blood pressure before versus after confinement | 3 months
Characterize clusters (homogeneous groups of patients) associated with particular dynamics of weight kinetics during confinement | 3 months
Evaluate the impact of teleconsultation monitoring during containment on weight loss | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, Principal Investigator — University Hospital, Grenoble
Locations (1):
- CHU Grenoble Alpes, Grenoble, France

REFERENCES:
- [Result] Bailly S, Fabre O, Legrand R, Pantagis L, Mendelson M, Terrail R, Tamisier R, Astrup A, Clement K, Pepin JL. The Impact of the COVID-19 Lockdown on Weight Loss and Body Composition in Subjects with Overweight and Obesity Participating in a Nationwide Weight-Loss Program: Impact of a Remote Consultation Follow-Up-The CO-RNPC Study. Nutrients. 2021 Jun 23;13(7):2152. doi: 10.3390/nu13072152. PMID 34201490